CLINICAL TRIAL: NCT02137096
Title: High Dose Conditioning With Ifosfamide, Carboplatin, and Etoposide With Autologous Stem Cell Transplantation for Patients With Recurrent Nasopharyngeal Carcinoma
Brief Title: Autologous Stem Cell Transplantation for Patients With Recurrent Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This is a rare disease, and enrollment was poor.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400316; PEDS008 (Other: University of Florida)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Nasopharynx Carcinoma
Keywords: Recurrent nasopharynx carcinoma
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — etoposide phosphate; Etoposide; Carboplatin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Dose Conditioning (Experimental): Single arm - receives high dose Etoposide phosphate, Ifosfamide, and Carboplatin followed by Autologous Stem Cell Transplantation
  Interventions: Drug: Etoposide phosphate; Drug: Carboplatin; Drug: Ifosfamide; Procedure: Autologous Stem Cell Transplantation

INTERVENTIONS:
Drug: Etoposide phosphate — Etoposide is one of three drugs used in the high-dose conditioning phase
  Other Names: Etopophos; Toposar
Drug: Carboplatin — Carboplatin is one of the drugs used in the high-dose conditioning phase.
  Other Names: Paraplatin
Drug: Ifosfamide — Ifosfamide is one of the drugs used in the high-dose conditioning phase
  Other Names: Ifex
Procedure: Autologous Stem Cell Transplantation — Autologous Stem Cell Transplantation follows the high-dose chemotherapy phase of the arm.

SUMMARY:
This is a pilot study to evaluate the response rates for patients undergoing high dose conditioning chemotherapy using Etoposide, Carboplatin and Ifosfamide followed by autologous stem cell transplantation for the treatment of recurrent Nasopharyngeal Cancer (NPC) in children, adolescents, and young adults.

DETAILED DESCRIPTION:
The use of high dose chemotherapy followed by autologous peripheral blood stem cell (PBSC) transplantation in recurrent nasopharyngeal carcinoma has shown promise when compared with standard chemotherapy. This study has been designed to evaluate response rates and toxicities associated with undergoing high dose conditioning with Etoposide, Carboplatin and Ifosfamide followed by autologous stem cell transplantation support in the treatment of recurrent nasopharyngeal carcinoma in children, adolescents, and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Imaging and tissue diagnosis of recurrent or progressive nasopharyngeal carcinoma
* Documentation of previous treatment including conventional chemotherapy and/or radiation therapy as clinically appropriate
* Ages 2 to 30 years of age
* Negative serum pregnancy test if applicable
* Calculated creatinine clearance of greater than 60 mL/minute, serum creatinine of less than 12o micromoles/L, total bilirubin less than 2 mg/dL and aspartate aminotransferase (AST) must be less than twice the upper limit of normal

Exclusion Criteria:

* Unsuitable candidate for autologous transplantation due to comorbidities or intractable psychosocial issues
* Pregnancy
* Breast-feeding women

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fort, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was terminated due to poor enrollment.
Period: Overall Study
Arm/Group | High Dose Conditioning
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High Dose Conditioning
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Tumor Response
Description: To evaluate the response rates for patients undergoing high dose conditioning using Etoposide, Carboplatin and Ifosfamide followed by autologous stem cell transplantation for the treatment of recurrent NPC in children, adolescents, and young adults.
Time Frame: 12 months after completion of treatment
Population: Due to only one subject being enrolled data analysis was completed
Arm/Group | High Dose Conditioning
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | High Dose Conditioning
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Conditioning (N=1)
Grade III Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Grade III Mucositis (Gastrointestinal disorders) | 1 (1)
Sepsis (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to no subject data analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT02137096/Prot_SAP_000.pdf